CLINICAL TRIAL: NCT00663351
Title: Post Approval Study: Reflection Ceramic Acetabular System
Brief Title: Safety and Effectiveness Study of the Reflection Ceramic Acetabular System
Acronym: RCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMA 030022
Record Dates: First submitted 2008-02-28; First posted 2008-04-22 (Estimated); Results first posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2015-03

CONDITIONS: Osteoarthritis
Keywords: Arthritis; Osteoarthritis; Traumatic Arthritis; Degenerative Joint Disease; Avascular Necrosis
MeSH Terms: conditions — Osteoarthritis; Arthritis; Joint Diseases; Osteonecrosis | interventions — Arthroplasty, Replacement, Hip

ARMS (2):
- Reflection Ceramic-Ceramic Hip System (IP) (Active Comparator): Investigational: Reflection Ceramic-Ceramic Hip System. Ceramic femoral head component and the ceramic acetabular cup insert are composed of Biolox forte aluminum oxide material.
  Interventions: Device: Reflection Ceramic-Ceramic Total Hip Replacement
- Reflection FSO V (5 hole) (Control) (Active Comparator): Control: Reflection FSO V (5 hole). Acetabular shell with a ultra high molecular weight polyethylene insert and an alumina ceramic femoral head with a Synergy or Spectron EF femoral stem. The Synergy femoral stem are composed of implant grade titanium while the Spectron EF stem is composed of implant grade cobalt chrome.
  Interventions: Device: Reflection FSO V Total Hip Replacement

INTERVENTIONS:
Device: Reflection Ceramic-Ceramic Total Hip Replacement — Intervention: all patients in study required (intervention) a total hip replacement, and were randomized to receive either the (Study Device)Reflection Ceramic Acetabular System or the(Control Device) Reflection FSO V (5 hole)acetabular system. Both arms received either a Synergy porous coated or Spectron EF stem.
  Other Names: Hip Replacement; Reflection; ceramic-ceramic
  Arms: Reflection Ceramic-Ceramic Hip System (IP)
Device: Reflection FSO V Total Hip Replacement — Intervention: all patients in study required (intervention) a total hip replacement, and were randomized to receive either the (Study Device)Reflection Ceramic Acetabular System or the(Control Device) Reflection FSO V (5 hole)acetabular system. Both arms received either a Synergy porous coated or Spectron EF stem.
  Other Names: Hip replacement; Reflection; ceramic-poly
  Arms: Reflection FSO V (5 hole) (Control)

SUMMARY:
This Post-Approval study is prospective follow-up study designed to evaluate the long-term safety and effectiveness of the Reflection Ceramic Acetabular System.

DETAILED DESCRIPTION:
This Post-Approval study is prospective follow-up study designed to evaluate the long-term safety and effectiveness of the Reflection Ceramic Acetabular System. Randomized Non-inflammatory Arthritis, Randomized Inflammatory and Continued Access Cohorts patients previously enrolled in the IDE study will be evaluated annually through five (5) year follow-up. In addition, all patients enrolled in the original study cohorts as well as the continued access patients will be sent a letter questionnaire annually at the 6-10 year postoperative time point to assess the patient's general well-being and if the study components are still in place

ELIGIBILITY:
Criteria

Inclusion Criteria:

(Patient must meet all of the following characteristics to be enrolled in the study):

* Males and females, 21 to 80 years of age, inclusive;
* Primary diagnosis of non-inflammatory arthritis (osteoarthritis) or inflammatory arthritis (rheumatoid arthritis), or patients requiring a revision as specified previously;
* The patient or his/her legal guardian is willing to consent to participate in the study by signing and dating the approved consent form;
* The patient will be available for follow-up through at least two years postoperative;
* The patient has met an acceptable preoperative medical clearance and is free or treated for cardiac, pulmonary, hematological, etc., conditions that would pose excessive operative risk (FDA requirement);
* The patient has a total Harris Hip Score of less than or equal to 60 (FDA requirement);
* The patient meets none of the exclusion criteria.

Exclusion Criteria:

(Patient with any of the following characteristics must be excluded from the study):

* Patients known to have insufficient quantity or quality of bone support resulting from Conditions such as cancer, femoral osteotomy, Girdlestone resection, significant osteoporosis or metabolic disorders of calcified tissues. Patients with physical conditions tending to place extreme loads on implants such as morbid obesity (> 100 pounds over desirable body weight), Charcot joints, muscle deficiencies, or multiple joint disabilities;
* Patients with active localized or systemic infection;
* Patients who have not reached full skeletal maturity;
* Patient psychological or neurological conditions which tend to preempt the patient's ability or willingness to restrict activities or follow medical advice, especially during the postoperative period, e.g.: drug or alcohol abuse, serious mental illness or retardation, or general neurological conditions;
* The patient is participating in any other pharmaceutical, biologic or medical device clinical investigation;
* Immunosuppressive disorders - immunosuppressive disorders are chronic conditions characterized by markedly inhibited ability to respond to antigenic stimuli. Examples of such conditions include patients who are on immunosuppressive therapy (corticosteroid hormones in large amounts, cytotoxic drugs, antilymphocytic serum or irradiation in large doses), patients receiving therapy to prevent homograft rejection, patients who have acquired immunodeficiency syndrome (AIDS), or auto-immune diseases (except rheumatoid arthritis).
* Pregnancy.
* Patients with known sensitivity to materials in the device.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2004-12; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Corpe, M.D., Principal Investigator — Medical College of Georgia, Dept of Orthopaedic; Joseph Zuckerman, M.D., Principal Investigator — Hospital of Joint Disease, Orthopaedic Institute; Jonathan P Garino, M.D., Principal Investigator — Presbyterian Medical Center, Dept of Orthopaedic; Michael J Grecula, M.D., Principal Investigator — University of Texas Medical Branch, Dept of Orthopaedic; James Howe, M.D., Principal Investigator — University of Vermont; Michael Lynch, M.D., Principal Investigator — The Memphis Orthopaedic Group, PC; Norman E Walter, M.D., Principal Investigator — Family Orthopaedics
Locations (7):
- United States (7):
  - Medical College of Georgia, Department of Orthopaedics, Augusta, Georgia
  - Family Orthopaedics, Flint, Michigan
  - Hospital of Joint Disease, Orthopaedic Institute, New York, New York
  - Presbyterian Medical Center, Department of Orthopaedic Surgery, Philadelphia, Pennsylvania
  - The Memphis Orthopaedic Group, PC, Memphis, Tennessee
  - University of Texas Medical Branch, Dept of Orthopaedics and Rehab, Galveston, Texas
  - University of Vermont College of Medicine, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 456 subjects (535 hips) enrolled initially at the beginning of the study. For the Post-Approval Study period (Year 6 through Year 10), 29 subjects (10 from the IP group, 19 from the control group) were excluded from analysis in the Intent-to-Treat (ITT) population and thus not included in the Participant Flow or Outcome Measures for this period.
Units Other Than Participants: Hips
Period: Initial Study (Year 1 up to Year 6)
Arm/Group | Reflection Ceramic-Ceramic Hip System (IP) | Reflection FSO V (5 Hole) (Control)
Started | 308; 372 Hips | 148; 163 Hips
Completed | 298; 364 Hips | 129; 144 Hips
Not Completed | 10; 8 Hips | 19; 19 Hips
Not completed — Lost to Follow-up | 10 | 19
Period: Post-Approval Study (Year 6 to Year 10)
Arm/Group | Reflection Ceramic-Ceramic Hip System (IP) | Reflection FSO V (5 Hole) (Control)
Started | 298; 364 Hips | 129; 144 Hips
Completed | 186; 252 Hips | 58; 73 Hips
Not Completed | 112; 112 Hips | 71; 71 Hips
Not completed — Revision Surgery | 29 | 10
Not completed — Withdrawal by Subject | 8 | 15
Not completed — Death | 18 | 7
Not completed — Lost to Follow-up | 13 | 7
Not completed — Withdrawn for Site Termination | 44 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reflection Ceramic-Ceramic Hip System (IP) | Reflection FSO V (5 Hole) (Control) | Total
Number analyzed (Participants) | 308 | 148 | 456
Age, Customized [Mean (Standard Deviation); unit: Years] | 48.7 (11.98) | 54.1 (12.91) | 50.7 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 71 | 218
  Male | 161 | 77 | 238
Height [Mean (Standard Deviation); unit: cm] | 173.0 (10.08) | 172.3 (9.83) | 172.7 (9.98)
Weight [Mean (Standard Deviation); unit: kg] | 86.4 (19.28) | 83.3 (18.78) | 85.3 (19.13)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (5.37) | 27.9 (5.14) | 28.4 (5.30)
Previous surgery on affected hip [Count of Participants; unit: Participants]
  Yes | 73 | 30 | 103
  No | 235 | 118 | 353
Other joint involvement [Count of Participants; unit: Participants]
  Yes | 216 | 99 | 315
  No | 92 | 49 | 141
Physical activity [Count of Participants; unit: Participants]
  None | 22 | 5 | 27
  Light | 225 | 113 | 338
  Moderate | 56 | 24 | 80
  Intense | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Survival of Hip Implant Based on Number of Hips Requiring Revision
Description: Revisions were assessed cumulatively from Initial Study Period through Post-Approval Study Period and End of Study/Withdrawal. Implant survival was analyzed based on the number of hip revisions that occurred as well as the cohort for each study arm (IP and Control), but further categorized by cohorts within each arm:
  RNIA = randomized, non-inflammatory arthritis cohort (IP or Control) RIA = randomized, inflammatory arthritis cohort (IP or Control) RR = revision cohort (IP or Control) CAC = continued access cohort (IP only)
Time Frame: Postoperatively through Year 10
Population: All hips/participants were assessed using the ITT population, which excluded 29 enrolled participants from analysis not meeting ITT criteria.
Measure: Count of Units; unit: Hips
Units Other Than Participants: Hips
Arm/Group | Reflection Ceramic-Ceramic Hip System (IP) | Reflection FSO V (5 Hole) (Control)
Number analyzed (Participants) | 298 | 129
Number analyzed (Hips) | 364 | 144
Hips
  Hips Requiring Revision: number analyzed (Hips) | 29 | 10
  Hips Requiring Revision: RNIA Cohort | 12 | 9
  Hips Requiring Revision: RIA Cohort | 2 | 1
  Hips Requiring Revision: RR Cohort | 0 | 0
  Hips Requiring Revision: CAC Cohort | 15 | 0
  Hips Not Requiring Revision: number analyzed (Hips) | 335 | 134
  Hips Not Requiring Revision: RNIA Cohort | 156 | 118
  Hips Not Requiring Revision: RIA Cohort | 17 | 9
  Hips Not Requiring Revision: RR Cohort | 5 | 7
  Hips Not Requiring Revision: CAC Cohort | 157 | 0

2. Primary Outcome: Survival of Hip Implant Based on Time Until Revision Required
Description: The survival of the implant was analyzed based on the length of time postoperatively until hip revision surgery was required (cumulatively through Initial Study Period and Post-Approval Study Period) for participants who required a revision surgery during the course of the study.
  The study arms were further categorized by cohorts within each arm:
  RNIA = randomized, non-inflammatory arthritis cohort (IP or Control) RIA = randomized, inflammatory arthritis cohort (IP or Control) RR = revision cohort (IP or Control) CAC = continued access cohort (IP only)
Time Frame: Postoperatively through Year 10
Population: Analysis is presented by individual hip ID numbers to demonstrate time before a revision was required as well as the corresponding cohorts of each. All hips/participants were assessed using the ITT population, which excluded 29 enrolled participants from analysis not meeting ITT criteria.
Measure: Number; unit: survival time in years
Units Other Than Participants: Hips
Arm/Group | Reflection Ceramic-Ceramic Hip System (IP) | Reflection FSO V (5 Hole) (Control)
Number analyzed (Participants) | 29 | 10
Number analyzed (Hips) | 29 | 10
survival time in years
  Hip ID 168 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 168 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 168 (RNIA cohort) | 0.0 |
  Hip ID 239 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 239 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 239 (RNIA cohort) |  | 0.0
  Hip ID 318 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 318 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 318 (RNIA cohort) |  | 0.0
  Hip ID 221 (RIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 221 (RIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 221 (RIA cohort) | 0.0 |
  Hip ID 348 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 348 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 348 (CAC cohort) | 0.0 |
  Hip ID 408 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 408 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 408 (CAC cohort) | 0.0 |
  Hip ID 448 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 448 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 448 (CAC cohort) | 0.0 |
  Hip ID 113 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 113 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 113 (RNIA cohort) | 0.1 |
  Hip ID 247 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 247 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 247 (RNIA cohort) | 0.1 |
  Hip ID 195 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 195 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 195 (RNIA cohort) | 0.3 |
  Hip ID 218 (RIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 218 (RIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 218 (RIA cohort) | 0.3 |
  Hip ID 458 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 458 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 458 (CAC cohort) | 0.3 |
  Hip ID 370 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 370 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 370 (CAC cohort) | 0.4 |
  Hip ID 398 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 398 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 398 (CAC cohort) | 0.4 |
  Hip ID 471 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 471 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 471 (RNIA cohort) | 0.7 |
  Hip ID 500 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 500 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 500 (CAC cohort) | 1.1 |
  Hip ID 412 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 412 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 412 (CAC cohort) | 1.3 |
  Hip ID 127 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 127 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 127 (RNIA cohort) | 1.8 |
  Hip ID 175 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 175 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 175 (RNIA cohort) | 2.2 |
  Hip ID 204 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 204 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 204 (RNIA cohort) | 2.5 |
  Hip ID 392 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 392 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 392 (CAC cohort) | 3.3 |
  Hip ID 306 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 306 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 306 (RNIA cohort) | 3.4 |
  Hip ID 483 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 483 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 483 (RNIA cohort) | 3.9 |
  Hip ID 167 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 167 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 167 (RNIA cohort) | 4.1 |
  Hip ID 451 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 451 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 451 (CAC cohort) | 4.2 |
  Hip ID 490 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 490 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 490 (CAC cohort) | 4.2 |
  Hip ID 288 (RR cohort): number analyzed (Participants) | 0 | 1
  Hip ID 288 (RR cohort): number analyzed (Hips) | 0 | 1
  Hip ID 288 (RR cohort) |  | 4.5
  Hip ID 37 (RNIA cohort): number analyzed (Participants) | 1 | 0
  Hip ID 37 (RNIA cohort): number analyzed (Hips) | 1 | 0
  Hip ID 37 (RNIA cohort) | 5.5 |
  Hip ID 110 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 110 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 110 (RNIA cohort) |  | 6.2
  Hip ID 337 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 337 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 337 (RNIA cohort) |  | 6.5
  Hip ID 496 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 496 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 496 (CAC cohort) | 6.8 |
  Hip ID 114 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 114 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 114 (RNIA cohort) |  | 6.9
  Hip ID 308 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 308 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 308 (RNIA cohort) |  | 7.0
  Hip ID 36 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 36 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 36 (RNIA cohort) |  | 7.9
  Hip ID 103 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 103 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 103 (RNIA cohort) |  | 7.9
  Hip ID 390 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 390 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 390 (CAC cohort) | 8.3 |
  Hip ID 385 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 385 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 385 (CAC cohort) | 8.4 |
  Hip ID 42 (RNIA cohort): number analyzed (Participants) | 0 | 1
  Hip ID 42 (RNIA cohort): number analyzed (Hips) | 0 | 1
  Hip ID 42 (RNIA cohort) |  | 8.9
  Hip ID 450 (CAC cohort): number analyzed (Participants) | 1 | 0
  Hip ID 450 (CAC cohort): number analyzed (Hips) | 1 | 0
  Hip ID 450 (CAC cohort) | 9.9 |

3. Primary Outcome: Subject Satisfaction Questionnaire
Description: A subject satisfaction questionnaire was conducted at Year 6, Year 7, Year 8, Year 9, and Year 10 postoperatively. The questionnaire was mailed to enrolled subjects each year (Years 6-10).
  The question was asked "Are you satisfied with hip?" and subjects responded either "yes" or "no".
Time Frame: Year 6 through Year 10 postoperatively
Population: The number analyzed include all enrolled subjects who responded to the questionnaire at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Reflection Ceramic-Ceramic Hip System (IP) | Reflection FSO V (5 Hole) (Control)
Number analyzed (Participants) | 298 | 129
Participants
  Year 6 - "Are you satisfied with hip?": number analyzed (Participants) | 110 | 25
  Year 6 - "Are you satisfied with hip?": Yes | 107 | 25
  Year 6 - "Are you satisfied with hip?": No | 3 | 0
  Year 7 - "Are you satisfied with hip?": number analyzed (Participants) | 190 | 51
  Year 7 - "Are you satisfied with hip?": Yes | 179 | 47
  Year 7 - "Are you satisfied with hip?": No | 11 | 4
  Year 8 - "Are you satisfied with hip?": number analyzed (Participants) | 194 | 48
  Year 8 - "Are you satisfied with hip?": Yes | 177 | 45
  Year 8 - "Are you satisfied with hip?": No | 17 | 3
  Year 9 - "Are you satisfied with hip?": number analyzed (Participants) | 208 | 50
  Year 9 - "Are you satisfied with hip?": Yes | 189 | 49
  Year 9 - "Are you satisfied with hip?": No | 19 | 1
  Year 10 - "Are you satisfied with hip?": number analyzed (Participants) | 224 | 60
  Year 10 - "Are you satisfied with hip?": Yes | 206 | 56
  Year 10 - "Are you satisfied with hip?": No | 18 | 4

ADVERSE EVENTS:
Time Frame: AEs were collected from enrollment through the end of the study/subject withdrawal whichever came first (up to 10 years). However, after the 5-year study report was presented to the FDA, only subject deaths were collected for AEs. The 6-10 year study requirement from the FDA included revision information, deaths, and subject satisfaction collection only.
Arm/Group | Reflection Ceramic-Ceramic Hip System (IP) | Reflection FSO V (5 Hole) (Control)
All-Cause Mortality (participants affected / at risk) | 18/308 | 7/148
Serious Adverse Events (participants affected / at risk) | 18/308 | 7/148
Other Adverse Events (participants affected / at risk) | 0/308 | 0/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reflection Ceramic-Ceramic Hip System (IP) (N=308) | Reflection FSO V (5 Hole) (Control) (N=148)
Complications related to an infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Injuries sustained during a house fire (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Found during a death index search, reason unknown (General disorders) | 3 (3) | 0 (0)
Unknown, not reported by site (General disorders) | 10 (10) | 3 (3)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats determined during the course of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No